CLINICAL TRIAL: NCT04897425
Title: Mindful SensoriMotor Therapy With Brain Modulation for the Treatment of Pain in Individuals With Disarticulation or Nerve Injuries: A Single Arm Clinical Trial
Brief Title: Mindful SensoriMotor Therapy With Brain Modulation in Highly Impaired Extremities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chalmers University of Technology (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Max Ortiz Catalan, Associate Professor, Chalmers University of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-07147
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Neuropathic Pain; Phantom Limb Pain
Keywords: Guided Plasticity therapy; Phantom Motor Execution; Mindful SensoriMotor Therapy; Brain Modulation; transcranial Direct Current Stimulation (tDCS); Neurological disorders; Neurobehavioral Manifestations
MeSH Terms: conditions — Neuralgia; Phantom Limb; Nervous System Diseases; Neurobehavioral Manifestations

STUDY DESIGN:
Intervention Model Description: Single arm clinical trial
Masking Description: However, the person treating the subject is different than the person evaluating the outcomes. This is done to reduce the influence that the care provider might have on the patient reporting positive outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful SensoriMotor Therapy Enhanced with Brain Modulation (Experimental): The participant can choose between one, two, or five interventions per week depending on their availability.
  Steps of each intervention:
  1. Pain Evaluation: Numeric Rating Scale (NRS)
  2. Functional Assessments (1st, 5th, 10th, and last sessions)
  3. Preparation:
     1. Locate participant in a comfortable position for training (comfortable chair, about a meter distance to the screen, pleasant arm position)
     2. Placement of the surface electrodes
     3. Positioning of the feedback wearable device over the affected body part
     4. Placement of the brain modulation cap
  4. Treatment modalities:
     1. Motor training
     2. Sensory training
     3. Sensorimotor training
  5. Assessments
  Step 4 is repeated for different phantom movements, initially one at a time, progressing to several joints simultaneously. A treatment session lasts 2 hours.
  Interventions: Device: Mindful SensoriMotor Therapy Enhanced with Brain Modulation

INTERVENTIONS:
Device: Mindful SensoriMotor Therapy Enhanced with Brain Modulation — Hardware and software for myoelectric pattern recognition and sensory training developed at the Center for Bionics and Pain Research.
  tES by Neuroelectrics

SUMMARY:
Brief summary: This single-arm, pilot clinical investigation aims to evaluate Mindful SensoriMotor Therapy (MSMT) enhanced with brain modulation as a treatment of pain due to sensorimotor impairment, such as Phantom Limb Pain (PLP). MSMT consists of consciously retraining the motor and sensory networks used by the missing limb via myoelectric pattern recognition and haptic feedback. In this trial, we further enhance the effect of MSMT by brain modulation, transcranial Direct Current Stimulation (tDCS).

DETAILED DESCRIPTION:
People with upper or lower limb disarticulation (amputation at joint level) or nerve injury will participate in this study. It is a single-arm study in which all participants receive the same intervention. Each participant attends a screening visit, up to 5 baseline assessments, 15 interventions, and 3 follow-ups at 1, 3, and 6 months after the last intervention. Brain imaging will be performed pre- and post-treatment.

ELIGIBILITY:
Inclusion criteria

* The participant has given written informed consent to participate.
* The participant must have chronic neuropathic pain due to sensorimotor impairment (example PLP).
* At least six months should be passed since the date of injury (acute pain cases should not be included in the study).
* If the participant is under pharmacological treatments, there must be no variations on the medication dosages (steady consumption) for at least 1 month before the screening visit.
* If the participant has previously been treated for neuropathic pain, the last session of that treatment(s) must be at least 3 months before the screening visit.
* Any pain reduction potentially correlated to previous neuropathic pain treatments must have been observed at least 3 months prior to the screening visit, as reported by the participant.
* In the case of having a prosthesis, the participant must be in a stable prosthetic situation (i.e. satisfied with the fitting of the prosthesis or not using a prosthesis).
* Participants must have enough contact surface at the site of the amputation or the injured nerves for the system to work, in the researcher's opinion.
* Participants must be able to perceive the haptic stimulation at the time of the screening visit.
* Participants must not experience painful sensations from haptic stimulation in the stump (i.e. allodynia).
* The participant has a sufficient understanding of both Swedish and English to be able to participate in all study assessments, in the researcher's opinion.
* Participants should not have any other condition or symptoms that can prevent them from participating in the study, in the researcher's opinion.
* No mental inability, reluctance, or language difficulties that result in difficulty understanding the meaning of study participation, in the researcher's opinion.
* The participant should not have any condition associated with the risk of poor protocol compliance, in the researcher's opinion.

Exclusion criteria

- The potential participant will be excluded from the study if the person does not meet at least one of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
The change in Pain Rating Index (PRI) over the treatment duration | Pain Rating Index registered at the beginning and at the end of the treatment. [ Time Frame: 28-40 weeks, depending on the frequency of the sessions.]
  The Pain Rating Index (PRI) is calculated as the sum of 15 descriptors presented to the participant at the end of each intervention session. Descriptors are rated from 0 (no pain) to 3 (maximum pain) and therefore, the PRI is a number between 0 and 45. The higher PRI number, the greater pain the person feels

SECONDARY OUTCOMES:
The change in Pain Disability Index (PDI) between the first and the last treatment session. | PDI assessed at the beginning the end of the treatment. [ Time Frame: 28-40 weeks, depending on the frequency of the sessions.]
  The Pain Disability Index (PDI) measures the impact of the pain on the ability of a person to participate in essential life activities. The PDI is the sum of 7 categories and each of the category rates between 0 and 10. Therefore, the index is comprised between 0 and 70. The higher the index the greater the person's disability due to pain is.

CONTACTS AND LOCATIONS:
Overall Officials: Max Ortiz Catalan, PhD, Principal Investigator — Associate Professor
Locations (1):
- Center for Bionics and Pain Research, CBPR, Mölndal, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The study protocol article will be published in a scientific journal.
Supporting Information: Study Protocol
Time Frame: The study protocol is estimated to be available from November 2021.
Access Criteria: open access

REFERENCES:
- [Background] Ortiz-Catalan M, Guethmundsdottir RA, Kristoffersen MB, Zepeda-Echavarria A, Caine-Winterberger K, Kulbacka-Ortiz K, Widehammar C, Eriksson K, Stockselius A, Ragno C, Pihlar Z, Burger H, Hermansson L. Phantom motor execution facilitated by machine learning and augmented reality as treatment for phantom limb pain: a single group, clinical trial in patients with chronic intractable phantom limb pain. Lancet. 2016 Dec 10;388(10062):2885-2894. doi: 10.1016/S0140-6736(16)31598-7. Epub 2016 Dec 2. PMID 27916234
- [Background] Lendaro E, Hermansson L, Burger H, Van der Sluis CK, McGuire BE, Pilch M, Bunketorp-Kall L, Kulbacka-Ortiz K, Rigner I, Stockselius A, Gudmundson L, Widehammar C, Hill W, Geers S, Ortiz-Catalan M. Phantom motor execution as a treatment for phantom limb pain: protocol of an international, double-blind, randomised controlled clinical trial. BMJ Open. 2018 Jul 16;8(7):e021039. doi: 10.1136/bmjopen-2017-021039. PMID 30012784
- [Background] Ortiz-Catalan M. The Stochastic Entanglement and Phantom Motor Execution Hypotheses: A Theoretical Framework for the Origin and Treatment of Phantom Limb Pain. Front Neurol. 2018 Sep 6;9:748. doi: 10.3389/fneur.2018.00748. eCollection 2018. PMID 30237784
- [Derived] Damercheli S, Buist M, Ortiz-Catalan M. Mindful SensoriMotor Therapy combined with brain modulation for the treatment of pain in individuals with disarticulation or nerve injuries: a single-arm clinical trial. BMJ Open. 2023 Jan 10;13(1):e059348. doi: 10.1136/bmjopen-2021-059348. PMID 36627156